CLINICAL TRIAL: NCT05553236
Title: Targeted Sequencing to Enhance, Liberate, and Optimize Treatment of Drug-resistant Tuberculosis
Brief Title: Pragmatic Use of Next-generation Sequencing for Management of Drug-resistant Tuberculosis
Acronym: TSELiOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Stellenbosch (Other); National Health Laboratory Service (NHLS), South Africa (Unknown); National Institute for Communicable Diseases, South Africa (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Find (Other); Translational Genomics Research Institute (Other); University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AI153213; R01AI153213 (NIH)
Record Dates: First submitted 2022-09-12; First posted 2022-09-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Drug-resistant Tuberculosis; HIV Coinfection; Cost-Benefit Analysis
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequencing Intervention in addition to standard of care (Experimental): Batched targeted deep sequencing in addition to the locally accepted standard of care drug susceptibility determination of multidrug/extensively drug-resistant tuberculosis (M/XDR-TB)
  Interventions: Diagnostic Test: Targeted next-generation sequencing
- Standard of Care (No Intervention): Locally accepted standard of care which is consistent with the WHO recommendations for the drug susceptibility determination of M/XDR-TB

INTERVENTIONS:
Diagnostic Test: Targeted next-generation sequencing — During intervention periods, an additional patient sample derived from routinely collected specimens will be processed by a local technician. Extracted DNA extracted from these samples will be batched on a regular basis for targeted deep sequencing. Sequencing results will be regularly transmitted to a clinical advisory committee.
  Arms: Sequencing Intervention in addition to standard of care

SUMMARY:
TS ELiOT is a stepped-wedge, cluster randomized trial assessing the effect of a next-generation sequencing-based strategy on rifampin-resistant tuberculosis management and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Active RR-TB diagnosed at a study facility during the study period
2. Positive Mtb culture, smear, or specimen derivative (e.g., GenoLyse remnant, Xpert cartridge extract)

Exclusion Criteria:

1. Patient expects to relocate/move residence outside of the study region
2. Patient does not agree to participate in the study

In addition, participants later found to have isolates with rifamycin susceptibility on at least two additional tests (e.g., phenotypic DST, LPA, or sequencing) will be considered late exclusions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with prespecified end of treatment outcomes | At the anticipated completion of prescribed treatment, up to 18 months
  The number of participants with each of the following prespecified end of treatment outcomes will be reported: cure, treatment completed, loss to follow up, treatment failure, death, transfer, and still on treatment.

SECONDARY OUTCOMES:
12-month relapse-free survival | From completion of prescribed treatment to death or TB recurrence, up to 12 months
  Length of time after treatment ends that the patient survives without TB recurrence
Exposure time to ineffective drugs | At the anticipated completion of prescribed treatment, up to 18 months
  Cumulative length of time on individual drugs to which Mtb is found to be resistant, per participant
Number of participants with acquired drug resistance | At the anticipated completion of prescribed treatment, up to 18 months
  Number of participants with M.tuberculosis acquiring additional drug resistance during treatment
Time to effective treatment initiation with three drugs | From diagnosis to treatment initiation with at least three effective drugs, up to 18 months
  Length of time from diagnosis to treatment initiation with at least three effective drugs to which M.tuberculosis is susceptible
Time to effective treatment initiation with four drugs | From diagnosis to treatment initiation with at least four effective drugs, up to 18 months
  Length of time from diagnosis to treatment initiation with at least four effective drugs to which M.tuberculosis is susceptible
Time to culture conversion | From diagnosis to stable culture conversion, up to 9 months
  Length of time from diagnosis to stable culture conversion, defined as the first of two (consecutive or non-consecutive) negative sputum cultures without an intervening positive culture, and/or visits wherein the participant is unable to produce sputum and has no signs of active TB, up to 9 months

OTHER OUTCOMES:
Number of participants with clinical uptake of sequencing intervention results | At the anticipated completion of prescribed treatment, up to 18 months
  The number of sequencing intervention results with treatment regimen adjustment where appropriate treatment change is indicated
Cost-effectiveness of the sequencing intervention | At the anticipated completion of prescribed treatment, up to 18 months
  Costs of necessary personnel, consumables, facility, logistics, and per unit tests

CONTACTS AND LOCATIONS:
Overall Officials: John Z Metcalfe, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- South African National Health Laboratory Service, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No